CLINICAL TRIAL: NCT06295640
Title: Relative Contribution of Brain Insulin Action for Postprandial Metabolism
Acronym: BrainInsPPM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Dr. med. Martin Heni, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 300/2022
Record Dates: First submitted 2024-02-08; First posted 2024-03-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Glucose Metabolism Disorders
Keywords: postprandial glucose metabolism; brain insulin action; insulin sensitivity; insulin secretion; endogenous glucose production; menstrual cycle; sex differences; proglucagon cleavage products
MeSH Terms: conditions — Glucose Metabolism Disorders; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cross-over design for men. Randomized, controlled, 2x2 factorial cross-over design for women taking the menstrual cycle phase into account.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal insulin spray (Experimental): 160 Units of human insulin as nasal spray
  Interventions: Other: Oral glucose tolerance test with double-tracer dilution and intranasal insulin spray
- Placebo spray (Placebo Comparator): Nasal spray containing placebo solution
  Interventions: Other: Oral glucose tolerance test with double-tracer dilution and intranasal placebo spray

INTERVENTIONS:
Other: Oral glucose tolerance test with double-tracer dilution and intranasal insulin spray — Subjects will undergo a 75 g OGTT (180 min) combined with a double tracer dilution. The double-tracer dilution technique will be used to quantify endogenous glucose production, glucose appearance and disappearance rate. [6,6-2H]glucose will be infused for a total of 300 minutes,while the infusion will start 120 minutes prior the OGTT and will last until the end of the OGTT. Intranasal insulin will be administered 15 minutes prior to the start of the OGTT. The drink consumed at time point 0 min contains 75 gram glucose, enriched with [U-13C6]-glucose.
  Arms: Intranasal insulin spray
Other: Oral glucose tolerance test with double-tracer dilution and intranasal placebo spray — Subjects will undergo a 75 g OGTT (180 min) combined with a double tracer dilution. The double-tracer dilution technique will be used to quantify endogenous glucose production, glucose appearance and disappearance rate. [6,6-2H]glucose will be infused for a total of 300 minutes,while the infusion will start 120 minutes prior the OGTT and will last until the end of the OGTT. Placebo spray will be administered 15 minutes prior to the start of the OGTT. The drink consumed at time point 0 min contains 75 gram glucose, enriched with [U-13C6]-glucose. To mimic insulin spill-over from nasal spray into systemic circulation, an i.v. insulin bolus of 3 mU × kg-1. will be administered over ten minutes starting at time point -15 minutes on the placebo spray day. On the insulin spray day a comparable amount of saline will be infused.
  Arms: Placebo spray

SUMMARY:
The goal of this clinical trial is to clarify (i) the contribution of brain insulin action on regulation of systemic metabolism, (ii) sex-specific differences in the central regulation and (iii) the influence of the menstrual cycle in women.

Therefore, participants will undergo oral glucose tolerance tests combined with a double tracer dilution technique. This approach will be compared between days with insulin delivery to the brain as nasal spray and days with placebo spray.

DETAILED DESCRIPTION:
This research project aims to investigate to what extent brain insulin action is responsible for the control of postprandial metabolism compared to direct effects of insulin in peripheral target tissues. Furthermore, the study will investigate sex differences and the influence of the menstrual cycle on brain-derived coordination of postprandial signaling for metabolic control.

Therefore, insulin action in the brain will be introduced by application of insulin as nasal spray (on one day) versus carrier solution as placebo nasal spray (on another day) in a randomized, blinded fashion. Spray administration will be performed 15 minutes before a 75 gram oral glucose tolerance test that will introduce a postprandial state. On placebo day, the known spillover of tiny amounts of nasal insulin into the systemic circulation will be mimicked by an appropriate i.v. insulin bolus. This approach will be combined with a double-tracer dilution technique. Labeled glucose ([6,6-2H]glucose) will be infused 120 minutes before and during the OGTT (180 min) and will be used to address endogenous glucose production. The glucose drink from the OGTT will be enriched with [U-13C6]glucose to compute the glucose appearance rate (Ra). Basal endogenous glucose production will be calculated as well as post-load endogenous glucose production and rates of glucose disappearances (Rd). Using this approach, brain-derived regulation of postprandial metabolism including endogenous glucose production, glucose disappearance, insulin secretion, and secretion of proglucagon-cleavage products (incretins) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 24 kg/m2
* no known primary diseases
* no hormonal contraception

Exclusion Criteria:

* Alcohol or drug abuse
* Smoking
* At screening: Hb < 12 g/dl for women and Hb < 14 g/dl for men
* Any (clinical) condition that would endanger participant's safety or question scientific success according to a physician's opinion.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Endogenous glucose production | -120 minutes - 180 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on endogenous glucose production assessed with Steele's non-steady state model during an oral glucose tolerance test combined with double-tracer dilution technique.
Rate of glucose disappearance | -120 minutes - 180 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on rate of glucose disappearance (Rd) assessed with Steele's non-steady state model during an oral glucose tolerance test combined with double-tracer dilution technique.

SECONDARY OUTCOMES:
Proglucagon cleavage products | 0-120 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on secretion of proglucagon cleavage products assessed by oral glucose tolerance test.
Glucose tolerance | 0-120 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on glucose tolerance assessed as area under the glucose curve (0-120 minutes) and glucose levels at timepoint 120 minutes during the 75 g oral glucose tolerance test.
Whole-body insulin sensitivity | 0-120 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on whole-body insulin sensitivity, assessed from glucose and insulin measurements during the 75 g OGTT.
Insulin secretion | 0-180 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on insulin secretion assessed from glucose and insulin/C-peptide measurements during the 75 g oral glucose tolerance test.
Post-absorptive energy expenditure | 30 minutes and 180 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on post-absorptive energy expenditure assessed by indirect calorimetry at timepoint 30 min and 180 min during an oral glucose tolerance test combined with double-tracer dilution technique.
Sex differences | -120 minutes - 180 minutes during oral glucose tolerance test
  Explore sex differences in the brain-derived regulation of postprandial metabolism during the 75 g oral glucose tolerance tests. Outcomes 1-7 will be compared between sexes.
Menstrual cycle effects | -120 minutes - 180 minutes during oral glucose tolerance test
  Differences between the follicular and the luteal phase of the menstrual cycle in the brain-derived regulation of postprandial metabolism during the 75 g oral glucose tolerance tests: Outcomes 1-7 will be compared between the phases of the menstrual cycle.
Autonomic nervous system activity | -15 minutes - 180 minutes during oral glucose tolerance test
  Effect of intranasal insulin versus placebo on autonomic nervous system activity assessed by heart rate variability using an 3-channel ECG at timepoint -15 min until 180 min during an oral glucose tolerance test combined with double-tracer dilution technique.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University of Ulm
Locations (1):
- Universityhospital Ulm, Ulm, Germany